CLINICAL TRIAL: NCT06759454
Title: Comparison of Mean Pain Score Using LASER Therapy and Desensitizing Agents in Patients With Dentinal Hypersensitivity: A Randomized Controlled Trial
Brief Title: Comparison of LASER Therapy and Desensitizing Agents in Dentinal Hypersensitivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kemia Gul (Other)
Responsible Party: Sponsor-Investigator, Kemia Gul, Comparison of Mean Pain Score Using Laser Therapy and Desensitizing Agents in Patients with Dentinal Hypersensitivity: A Randomized Controlled Trial, College of Physicians and Surgeons Pakistan
Organization: College of Physicians and Surgeons Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208-ERB/024
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Dentinal Hypersensitivity
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 (Desensitizing Agent) (Active Comparator): A glutaraldehyde-based desensitizing agent applied to affected teeth for 30 seconds, air-dried, with post-application instructions
  Interventions: Drug: Glutaraldehyde-Based Desensetizing Agent
- Arm 2 (Laser Therapy) (Experimental): Diode laser set to 100 mW in continuous wave mode, applied to specific areas of affected teeth for three minutes
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Drug: Glutaraldehyde-Based Desensetizing Agent — A glutaraldehyde-based desensitizing agent applied to the cervical area of affected teeth using a micro-brush, left undisturbed for 30 seconds, and air-dried. Both interventions aim to reduce pain associated with dentinal hypersensitivity by either occluding dentinal tubules or reducing nerve excitability
  Arms: Arm 1 (Desensitizing Agent)
Device: Low Level Laser Therapy — Low-level laser therapy (LLLT) using a diode laser set to a low power level (e.g., 100 mW, continuous wave mode). Each affected tooth will be treated for three minutes, targeting apical, cervical, and middle points
  Arms: Arm 2 (Laser Therapy)

SUMMARY:
This study evaluates the effectiveness of laser therapy versus desensitizing agents in reducing pain among participants with dentinal hypersensitivity conducted in Saidu College of Dentistry. Pain will be measured at baseline, immediately post-treatment, one week, and three months using the Visual Analog Scale (VAS)

DETAILED DESCRIPTION:
This study examines dentinal hypersensitivity treatment modalities, including laser therapy and desensitizing agents. The study is conducted in compliance with regional ethical guidelines

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-50 years with a preoperative VAS score of ≥2 for dentinal hypersensitivity.
* Participants with sensitivity due to gingival recession, cervical abrasion, or enamel erosion.
* Participants with good systemic health.
* Minimum of two hypersensitive teeth present in two different quadrants.

Exclusion Criteria:

* Teeth with caries, defective restorations, or cervical defects > 2 mm (may affect sensitivity measurements).
* Periodontal surgery or deep periodontal pockets (> 6 mm) within the past three months (potential influence on periodontal health and sensitivity).
* Participants using desensitizing toothpaste within the past three months (could interfere with study outcomes).
* Presence of gross oral pathology or systemic diseases (e.g., eating disorders, chronic diseases, uncontrolled metabolic conditions) (may alter oral health status).
* Pregnant or lactating women (hormonal changes can influence oral health).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity: Visual Analog Scale | Immediately post-treatment, one week, and three months
  After intervention there is a possibility of change in pain intensity in Dentinal Hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: BREKHNA YOUSAFZAI, Principal Investigator — Saidu College of Dentistry
Locations (1):
- Saidu College of Dentistry, Swat, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers due to confidentiality concerns, ethical considerations, and the absence of any formal plan for data sharing at this time